CLINICAL TRIAL: NCT06552611
Title: Non-invasive Electrical Spinal Cord Stimulation To Restore Upper Extremity Function in Multiple Sclerosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Sarah Simmons, MD, PhD, Assistant Professor, Department of Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00020787
Record Dates: First submitted 2024-08-08; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Multiple Sclerosis
Keywords: Rehabilitation; Neuromodulation; Spinal Cord stimulation
MeSH Terms: conditions — Multiple Sclerosis | interventions — Therapeutics; Occupational Therapy

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-label, two-intervention arm cross-over clinical trial of transcutaneous spinal cord stimulation combined with therapy compared to therapy alone in four adults with MS and upper extremity impairment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hand Therapy alone (Active Comparator): Participants randomized to hand therapy alone will participate in therapy sessions three times per week, 60 minutes per session for six weeks.
  Interventions: Other: Occupational Therapy
- Hand Therapy + Stimulation (Experimental): Participants will receive non-invasive transcutaneous electrical spinal cord stimulation paired with hand therapy sessions three times per week, 60 minutes per session, for six weeks.
  Interventions: Combination Product: Transcutaneous electrical spinal cord stimulation + therapy; Other: Occupational Therapy

INTERVENTIONS:
Combination Product: Transcutaneous electrical spinal cord stimulation + therapy — A two-channel transcutaneous spinal cord stimulator (SCONE, SpineX, Inc.) will deliver non-invasive electrical stimulation during hand therapy sessions. For each session, two self-adhesive hydrogel electrodes will be positioned along the midline of the C3-C4 and C6-C7 spinous processes over the skin as cathodes to stimulate the cervical spinal cord at two vertebral levels. An additional pair of electrodes will be symmetrically positioned over either the iliac crests or shoulders, functioning as anodes. The electrical current employed for the transcutaneous spinal cord stimulation is biphasic, featuring a 1-millisecond pulse width, a base frequency of 30 Hz, and an overlapping frequency of 10 kHz. Stimulation intensity will range from 0 to 120 milliamperes (mA), with incremental increases of 5 mA until reaching the level that facilitates voluntary movement. The stimulation amplitude will be fine-tuned for each specific activity based on the therapist's observation.
  Other Names: Open-loop stimulation
  Arms: Hand Therapy + Stimulation
Other: Occupational Therapy — The hand therapy program is comprised of intensive, progressive, functional task practice following a standardized protocol. The protocol consists of repetitive activities of gross upper limb movement, isolated finger movements, bimanual task performance, simple and complex pinch, and grip performance. Several activities with various difficulty levels are designated for each category, and the participant will perform 1-2 activities within each category in each training session. Activities are chosen according to the participant's ability, interests, and needs and are modified as function progresses over time.
  Other Names: hand therapy; functional task practice

SUMMARY:
Current disease-modifying therapies for multiple sclerosis (MS) aim to prevent the development of new lesions; unfortunately, no current FDA-approved therapies promote central nervous system (CNS) repair mechanisms. Thus, strategies to promote functional recovery from lesion-related deficits in adults with MS remain an unmet need.

This is a pilot study designed to test the feasibility, safety and preliminary efficacy of non-invasive (transcutaneous, applied by surface electrodes over the skin) electrical spinal cord stimulation combined with occupational therapy for restoring upper extremity sensorimotor function in adults with multiple sclerosis.

Participants with multiple sclerosis and impaired upper extremity function will complete two separate 6-week intervention sessions: 6 weeks of occupational therapy combined with transcutaneous spinal cord stimulation and 6 weeks of occupational therapy alone. The order of these interventions will be randomized, and each intervention will be separated by a 6-week washout period.

The investigators hypothesize that:

1. transcutaneous spinal cord stimulation combined with therapy will be feasible and acceptable by participants
2. transcutaneous spinal cord stimulation combined with therapy will lead to improvements in upper extremity function compared to occupational therapy alone
3. transcutaneous spinal cord stimulation combined with therapy will lead to improvements in symptoms related to quality of life (pain, spasticity, and bladder symptoms) compared to occupational therapy alone

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MS
2. Age between 21 and 70
3. Presence of upper extremity functional impairment (correlating with raw score ≤34 on NeuroQOL Upper Extremity Function short-form questionnaire),
4. Ability to attend intervention and assessment sessions 3 times per week.
5. For women of childbearing potential, willingness to provide confirmation of a negative over-the-counter home pregnancy test within 2 weeks of study entry and prior to each intervention arm.

Exclusion Criteria:

1. Relapse within the past 6 months (given that natural recovery from relapse could skew results)
2. Active implanted stimulator or baclofen pump
3. Upper extremity botox injection within the past 6 months
4. Unstable dalfampridine usage during study duration (which may interfere with functional outcomes)
5. Coexisting neurological condition that could interfere with interpretation of testing results (hx of stroke, traumatic brain injury, epilepsy/seizure, ALS, spinal cord injury, central nervous system vasculitis, intracranial tumor, intracranial aneurysm, cervical myelopathy/radiculopathy or peripheral neuropathy (diabetic polyneuropathy, entrapment neuropathy), etc.)
6. History of major active psychiatric illness that could interfere with treatment, such as severe depression, alcohol/drug abuse, or dementia
7. Serious comorbidities (e.g., cardiac arrhythmia, uncontrolled hypertension, respiratory disease, cancer, renal failure, chronic infectious disease, rheumatic disease, frequent UTIs, etc.) that would prevent participation in study activities
8. Presence of severe joint contractures in the affected hand and arm that may interfere with study activities or outcome measures
9. Severe spasticity, as defined by an Ashworth score of 4 in both sides of the upper limb
10. Pregnant and/or breastfeeding
11. Lack of ability to fully comprehend, cooperate, and/or safely perform study procedures in the investigator's opinion/judgment
12. Inability to give consent

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Nine-Hole Peg Test | 6 weeks
  Nine-Hole Peg Test is a standardized, quantitative assessment used to measure finger dexterity. Score is time it takes to complete task (range 15-180 seconds). Higher score = worse outcome.
NeuroQoL Upper Extremity Function | 6 weeks
  A self-report of health-related quality of life for adults with neurological disorders. Score ranges from 8-40; higher score = better function
Participant Drop-out rate | 6 weeks
  Percentage of participants who complete the intervention protocol. (0-100%)

SECONDARY OUTCOMES:
Action Research Arm Test | 6 weeks
  A 19-item clinician-administered observational measure to assess upper extremity performance (coordination, dexterity, and functioning). Items comprising the ARAT are categorized into four subscales (grasp: 6 items, score 0-18; grip: 4 items, score 0-12; pinch: 6 items, score 0-18; and gross movement: 3 items, score 0-9) and arranged in order of decreasing difficulty, with the most difficult task examined first, followed by the least difficult task. Scores are aggregated to a final scale (ranging from 0-57); Higher scores indicate better performance.
Box and Blocks Test | 6 weeks
  Measures unilateral gross manual dexterity. The test kit comprises a wooden box divided into two compartments by a partition and 150 blocks. Participants move, one by one, the maximum number of blocks from one compartment of a box to another of equal size within 60 seconds. Score ranges from 0-150; higher score indicates better function.
Grip force | 6 weeks
  measurement of hand strengths using dynamometry. Measured in pounds (score ranges from 0-200); higher score indicates better function.
Pinch force | 6 weeks
  measurement of hand strengths using dynamometry. Measured in pounds (score ranges from 0-100); higher score indicates better function.
Modified Ashworth Scale | 6 weeks
  A clinician-administered test for resistance of a joint to the passive movement. This scale grades the muscle tone from 0 (normal) to 4 (severe spasticity). Higher score indicates worse function
Patient-reported Impact of Spasticity Measure | 6 weeks
  A patient-reported outcome questionnaire assessing the impact of spasticity on function and quality of life over the past week. Score ranges from 0-164; higher scores indicate worse function.
Modified Fatigue Impact Scale | 6 weeks
  A patient-reported outcome questionnaire. It is a modified form of the Fatigue Impact Scale based on items derived from interviews with multiple sclerosis patients concerning how fatigue impacts their lives. This instrument provides an assessment of the effects of fatigue on physical, cognitive, and psychosocial functioning. Score ranges from 0-84; higher score indicates worse function.
PROMIS Pain Interference | 6 weeks
  A patient-reported outcome questionnaire that measures the self-reported consequences of pain on relevant aspects of a person's life and may include the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. Score ranges from 4-20; higher score indicates worse function.
PROMIS Pain Intensity | 6 weeks
  A patient-reported outcome numeric rating scale of pain over the past 7 days. Score ranges from0-10; higher score indicates worse pain
Bowel Control Scale | 6 weeks
  A patient-reported outcome questionnaire for bowel management. This is a subsection of the Multiple Sclerosis Quality of Life Inventory. Score ranges from 0-26; higher score indicates worse function.
Bladder Control Scale | 6 weeks
  A patient-reported outcome questionnaire for bladder management. This is a subsection of the Multiple Sclerosis Quality of Life Inventory. Score ranges from 0-22; higher score indicates worse function.
Global Impression of Change | 6 weeks
  A patient and clinician-reported scale of change pre- to post-intervention, ranging from 1 (indicating "very much improved") to 7 (indicating "very much worse").
Ability to Participate in Social Roles and Activities | 6 weeks
  A self-report of health-related quality of life in 17 domains and sub-domains for adults with neurological disorders. Score ranges from 4-40; higher scores indicates better function.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Simmons, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States